CLINICAL TRIAL: NCT04193722
Title: The Effect of Hyperbaric Oxygen Therapy on Breast Cancer Patients With Late Radiation Toxicity
Brief Title: The Effect of Hyperbaric OxygeN Therapy on brEast Cancer Patients With Late Radiation toxicitY - UMBRELLA HONEY Trial
Acronym: HONEY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Prof. dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL69081.041.19
Record Dates: First submitted 2019-11-11; First posted 2019-12-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Radiation Toxicity
Keywords: Breast cancer; Radiotherapy; Hyperbaric oxygen therapy; Late toxicity; Trials within cohorts; Patient reported outcomes
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries | interventions — Hyperbaric Oxygenation; Oxygen

STUDY DESIGN:
Intervention Model Description: Trial within cohorts design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric oxygen therapy (Experimental): Hyperbaric oxygen therapy consists of 30-40 treatment sessions (1 session per day during 5 days per week). During the hyperbaric oxygen (HBO) sessions the pressure will be raised to 2.4 atmospheres absolute in a hyperbaric chamber and patients breath in 100% oxygen during 4 times 20 minutes.
  Interventions: Drug: Hyperbaric oxygen therapy
- Usual care (No Intervention): Usual care may consist of physiotherapy, analgetics, edema therapy

INTERVENTIONS:
Drug: Hyperbaric oxygen therapy — Hyperbaric oxygen therapy in a multiperson hyperbaric oxygen chamber. Standard hyperbaric oxygen therapy provided as reimbursed by insurers.
  Other Names: Oxygen
  Arms: Hyperbaric oxygen therapy

SUMMARY:
The "Hyperbaric OxygeN therapy on brEast cancer patients with late radiation toxicity" (HONEY) trial aims to evaluate the effectiveness of HBOT on late radiation toxicity in breast cancer patients using the trial within cohorts (TwiCs) design.

DETAILED DESCRIPTION:
Objective: The aim of this study is to assess whether HBOT reduces pain, and improves physical functioning and QoL in breast cancer patients with late radiation toxicity.

Study design: Randomized controlled trial, nested within the prospective UMBRELLA breast cancer cohort according to the TWiC's design. UMBRELLA is a prospective cohort study including all breast cancer patients visiting the University Medical Center (UMC) Utrecht department of Radiotherapy. In total 120 patients will be randomized in a ratio of 2:1.

Study population: Breast cancer patients participating in the UMBRELLA cohort who have given informed consent to be invited for future research (e.g. cmRCT's), and who have reported symptoms of late radiation toxicity.

Intervention: Eligible patients will be referred to the HBO center for a standard HBO treatment. HBOT consists of 30-40 treatment sessions (1 session per day during 5 days per week). During the hyperbaric oxygen (HBO) sessions patients breath in 100% oxygen during 4 times 20 minutes in a hyperbaric chamber.

Main study parameters/endpoints: The primary endpoint of this study is patient reported breast/chest wall pain. Secondary endpoints are: physical functioning, QoL cosmetic outcome, physician reported pain and radiation toxicity (according to CTCAE criteria version 4.03, tissue oxygenation previous to HBOT and after HBOT and side-effects of HBOT.

ELIGIBILITY:
Inclusion Criteria:

* Self reported pain grade 3-4 (on a scale of 1-4) as assessed by the late radiation toxicity questionnaire;
* Participation >12 months in the UMBRELLA cohort;
* Previous treatment with radiotherapy for breast cancer;
* Completed surgery and (neo)adjuvant systemic therapy except adjuvant endocrine therapy, for breast cancer.

Exclusion Criteria:

* Poor responder to questionnaires (i.e. return of ≤ 2 UMBRELLA questionnaires);
* Previous HBOT;
* Contra-indications for HBOT (e.g. (severe) chronic obstructive pulmonary disease (COPD) or asthma, pacemaker, morbid obesity, epilepsy in medical history, severe heart failure);
* Current metastatic disease or recurrent breast cancer.

Additional exclusions criteria based on screening visit:

* Inability to follow schedule of all consecutive HBO treatments (e.g. due to scheduled holidays > 2 days);
* Not meeting criteria for HBOT (e.g. due to complaints similar to late radiation toxicity, not caused by radiotherapy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Change in breast/chest wall pain: EORTC QLQ-BR23 questionnaire | Baseline and 6 months after baseline (i.e. 3 months after HBOT)
  The primary endpoint of this study is the difference in proportion of patient-reported breast/chest wall pain grade 3-4 between control and intervention group. Pain is assessed by means of the EORTC QLQ-BR23 questionnaire on a 4-point Likert scale. At baseline all patients have a pain score of 3 or 4 (see inclusion criteria). The proportion of patients with 3-4 at 6 months will be compared between intervention and control group. A higher score indicates more pain.

SECONDARY OUTCOMES:
Change in patient-reported quality of life: (EORTC QLQ) C30 | Baseline and 6 months after baseline (i.e. 3 months after HBOT)
  Quality of life (QoL) measured by European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30. QoL will be scored on a scale of 0-100. A higher score indicates a better outcome. Change in score between baseline and 6 months will be compared between intervention and control group.
Change in patient-reported late radiation toxicity | Baseline and 6 months after baseline (i.e. 3 months after HBOT)
  Late radiation toxicity is assessed by means of a late radiation toxicity questionnaire (ability to move the arm, (breast) edema, fibrosis) in both control group and intervention group. Change in patient reported late radiation toxicity will be compared between intervention and control group. Late radiation toxicity will be assessed on a 4-point Likert scale. A higher score indicates worse outcomes.
Physician-reported late radiation toxicity | Baseline (prior to HBOT), 3 months after baseline (i.e. after HBOT) and 6 months after baseline (i.e. 3 months after the last HBO session)
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 only in intervention group. CTCAE criteria are assessed on a scale of 0-3.
Patient-reported cosmetic outcome | Baseline and 6 months after baseline (i.e. 3 months after HBOT)
  Assessed by means of the breast cancer questionnaire (BREAST-Q) in both control group and intervention group. BREAST-Q scores will be assessed using the BREAST-Q scoring tables.
Physician-reported cosmetic outcome | Baseline and 6 months after baseline (i.e. 3 months after HBOT)
  Reported by means of medical photograph (cosmetic outcome judged by group of experts and "Breast Cancer Conservative Treatment - cosmetic results" (BCCT.core) program) and with physical examination using the Patient and Observer Scar Assessment Scale (POSAS) score v2.0. Physician reported cosmetic outcome will only be assessed in the intervention group.
Number of participants with side effects of treatment with hyperbaric oxygen therapy | During hyperbaric oxygen treatment sessions and at 3 months after last HBO session
  Side effects of HBOT will be monitored using the MacFie classification only in the intervention group.
Oxygenation of the skin | Baseline and prior to last hyperbaric oxygen session (i.e. 3 months after baseline).
  Skin oxygenation will be measured prior to HBOT and after last treatment session using transcutaneous oxygen measurement. The contralateral breast will be used as a reference. Only assessed in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Helena M Verkooijen, MD, PhD, Principal Investigator — Imaging Division, UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Mink van der Molen DR, Batenburg MCT, Maarse W, van den Bongard DHJG, Doeksen A, de Lange MY, van der Pol CC, Evers DJ, Lansdorp CA, van der Laan J, van de Ven PM, van der Leij F, Verkooijen HM. Hyperbaric Oxygen Therapy and Late Local Toxic Effects in Patients With Irradiated Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2024 Apr 1;10(4):464-474. doi: 10.1001/jamaoncol.2023.6776. PMID 38329746
- [Derived] Batenburg MCT, van den Bongard HJGD, Kleynen CE, Maarse W, Witkamp A, Ernst M, Doeksen A, van Dalen T, Sier M, Schoenmaeckers EJP, Baas IO, Verkooijen HM. Assessing the effect of hyperbaric oxygen therapy in breast cancer patients with late radiation toxicity (HONEY trial): a trial protocol using a trial within a cohort design. Trials. 2020 Nov 27;21(1):980. doi: 10.1186/s13063-020-04869-z. PMID 33246494